CLINICAL TRIAL: NCT00154934
Title: The Impact of Interleukin-10 in the Invasion Capacity and Immunoregulation During Pregnancy: the Implications of Pathogenesis of Pre-Eclampsia.
Brief Title: the Implications of Pathogenesis of Pre-Eclampsia
Status: Terminated | Type: Observational
Why Stopped: difficult to enroll subjects
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 9361700215
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — placenta biopsy
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Preeclampsia is a severe complication of human pregnancy. It occurs in 4-5% of all pregnancies and remains a leading cause of maternal and neonatal mortality and morbidity. The pathophysiology of this syndrome is not fully understood. Two theories are proposed to explain the development of preeclampsia: defective trophoblast invasion in the first trimester, and poor maternal immunoregulation against the fetus. Pro-inflammatory cytokines are induced in the second mechanism, with a subsequent generalized endothelial dysfunction in the mother. Interleukin-10 (IL-10) plays a major role in this pathway.

According to recent literature, debates still exist on the role of IL-10 in the pathogenesis of preeclampsia. IL-10 may increase immunoregulation (seemingly against the development of preeclampsia), but also prohibit the extravillous trophoblast invasion on the other hand (seemingly towards the development of preeclampsia). According to recent authoritative journals, the expression of IL-10 pre-eclamptic placenta is increased; but some other influential journals have the totally contrary results. We believe this diverse exhibition may be due to overlook the paracrine effect of decidual cells (representative of maternal environment), and in vitro cultured condition does not parallel to physiological condition.

Our experiment has first obtained the qualification of Ethical Committee of our hospital and the permission of the examined patients. We first collect the serum sample of preeclampsia patient and analyze the IL-10 level by ELISA kit, and compared with normal control. Then we isolate trophoblast from pre-eclamptic women and normal control. These trophoblasts are further treated with (1) co-cultured with decidual cell line (2) Lipofectamine transfection with IL-10 (overexpression of IL-10) (3) signal interference ribonucleotide (siRNA) of IL-10 (knockdown IL-10 function). Each groups (including trophoblast alone from patients or normal control) were subjected to the analysis of IL-10 mRNA amount by RT-PCR. Further experiments for these treated trophoblast are transwell migration assay and invasion assay, matrix metalloproteinase assay to determine the change of invasive capacity; and Fas ligand expression to determine the change of immunoregulation.

Our effort is not only to determine the role of IL-10 in the pathogenesis of preeclampsia, but also the development of siRNA IL-10 may give a light in the treatment of preeclampsia.

DETAILED DESCRIPTION:
1. Pregnancy, pre-eclampsia and immune regulation The preeclampsia syndrome, which is characterized by changes in the placenta and uteroplacental vasculature, is a major concern in impaired human pregnancy. Hypertension, proteinuria and exaggerated edema are typical clinical symptoms1. Although the etiology of the disease is uncertain, it is well established that a defect in placental trophoblast invasion during implantation contributes to inadequate remodeling of uterine spiral arteries, thereby initiating focal regions of reduced perfusion within the placenta2. It has been suggested that a consequence of placental ischemia is the generation of cytotoxic factors that may act systemically to activate or injure the endothelium3. The identity of the factors elaborated by the placenta, which presumably compromise endothelial function during preeclampsia, is unknown. Inflammatory cytokines, such as tumor necrosis factor-α (TNF-α) and interleukin-1β (IL-1β), are known to be potent activators of the vascular endothelium and have been proposed as mediators of endothelial dysfunction during preeclampsia4.

   It is well known that the acceptance of the fetoplacental unit in human pregnancy requires maternal immune tolerance, which is thought to be regulated locally by the placenta. Therefore an anti-inflammatory cytokine, such as interleukin-10 plays a critical role in different pregnancy disorders, including preeclampsia5.

   Placental interleukins have been identified in reproductive tissues, but their roles in adaptive maternal immunity and determining term pregnancy outcomes have not been fully clarified. The acceptance of the fetoplacental unit by the maternal uterine surface requires an element of immunological tolerance. Local antiplacental immunity is modified by synthesis of uncommon histocompatibility Ags, growth factors, and cytokines by the placenta. The presence of immune cells in the decidual tissue of the uterus also presents a potential barrier, both physical and immunological, to the development of the placenta6. Some characteristics of the fetoplacental unit encourage endometrial and myometrial invasion7 and others modify the immunological barrier (e.g. HLA-G)8. These characteristics of placental function may be abnormal at the formative stages of placental development, and thus the presumptive uterine barriers may be abnormal in preeclampsia, a complication of human pregnancy related to shallow placental development9.
2. Interleukin-10 Interleukin-10 was originally identified as the product of Th2-type T lymphocytes that inhibits the synthesis of Th-1 type cytokines such as Interferon-gamma and IL-210. IL-10 is known to be secreted by Th2-helper T cells, CD4+HT2 cells, and some B cell lymphoma and mast cell lines. The protein undergoes post-translational modification that includes N-glycosylation and the formation of critical cysteine bonds. IL-10 inhibits cytokine synthesis in both T cells and NK cells by controlling macrophage-monocyte accessory cells. IL-10 elicits responses in granulocytes, eosinophils, mast cells, B cells, T cells and NK cells11. IL-10 is crucial in limiting inflammatory responses in some disease states. The ability of IL-10 to inhibit macrophage activation should allow investigation into "cross-talk" between stimulatory and inhibitory cytokines. IL-10 is important in understanding autoimmunity and as a target molecule in the development of anti-rejection therapies12. The Th-like responses of this cytokine make it a suitable adjuvant for immunization development10.

   Human and mouse IL-10 are 73% homologous at the amino acid level. Human IL-10 is active in mouse cell lines, but human cell lines are not responsive to mouse IL-10.
3. Maintenance of pregnancy and interleukin-10 production Interleukin-10 (IL-10) is an immunosuppressive cytokine expressed throughout pregnancy by epithelial cells and leukocytes in the endometrium and placenta. The anti-inflammatory and immune deviating properties of IL-10 are well characterized. Principally these are mediated through inhibiting proliferation and pro-inflammatory cytokine synthesis in type 1 T helper (Th1) cells, programming specific phenotypes in macrophages and dendritic cells and stimulating natural killer (NK) cell activation.

   IL-10 has been shown in normal placental cells (trophoblast cells) to suppress the mixed lymphocyte responses in vitro13. Maternal bone marrow-derived cells in the uterine wall include NK-like cells and T cells14 that may be modified by placental IL-10 production. Modification of the local maternal antifetal immune response has been shown to be important in patients with recurrent spontaneous abortion15.

   IL-10 has been identified as an important cytokine in pregnancy. IL-10 may be involved in the maintenance of pregnancy by corpus luteum maturation and progesterone production16. In a well-known mouse cross that is prone to spontaneous abortion a deficiency of IL-10 has been demonstrated to alter the net fetal number and outcome17. Longitudinal studies in mice demonstrate a sequential change in the cytokine profile including IL-10 in peripheral blood and release from spleen elements as pregnancy advances18,19. IL-10 inhibition in the second half of pregnancy in mice causes fetal growth retardation20. Besides, progesterone has been shown to increase Th2-type responses in T cells21. Taken together, these data suggest that early pregnancy is associated with an increase in circulating Th2 cytokine IL-10 and that fetal and placental growth and development are depend on adequate IL-10 production. Or in brief, IL-10 may have a fetal protective effect.

   In human pregnancy there is a shift of cytokine production from Th1-type inflammatory cytokines to Th2 type cytokines with a predominance of IL-10 and IL-4 over IL-2 and TNF-α in stimulated PBMC. This balance altered in preeclamptic mononuclear cells with the alternative result, a relative decrease in IL-10 compared with the pro-inflammatory cytokine production22.
4. Interleukin-10 on trophoblast motility and invasion capacity Interleukin-10, expressed in the decidua and placenta, is implicated in regulating extravillous cytotrophoblast invasion through inhibiting matrix metalloproteinase expression and influencing the quality of the maternal immune response.

   Cytotrophoblast invasion in vitro requires the expression of matrix metalloproteinase-9 (MMP-9). In a recent article, the authors showed that cytotrophoblasts produce interleukin-10 (IL-10), a potent immunomodulatory cytokine that could have paracrine effects on the maternal immune system. IL-10 synthesis is dramatically downregulated after the first 12 h of culture, while MMP-9 secretion is rapidly upregulated and the cells acquire an invasive phenotype.13 These observations prompted the subsequent experiments to investigate whether IL-10 is an autocrine regulator of cytotrophoblast MMP-9 production. Adding recombinant IL-10 to cytotrophoblast cultures significantly decreased the cells' MMP-9 expression at both protein and mRNA levels, but did not affect mRNA levels of the tissue inhibitor of metalloproteinase-3.23 Thus, IL-10 may alter the proteinase/inhibitor balance. IL-10 treatment further caused a net decrease in MMP activity, thereby reducing cytotrophoblast invasiveness. Together, the current data suggest that IL-10 is an autocrine inhibitor of cytotrophoblast MMP-9 activity and invasiveness.
5. Controversies of interleukin-10 and the development of preeclampsia Endothelial cell dysfunction has been hypothesized to be a major contributor in the pathogenesis of pre-eclampsia. This hypertensive disease of pregnancy is characterized by changes in the placenta, uteroplacental vasculature, kidneys, and liver consistent with endothelial damage. Hypertension and vascular hypersensitivity to pressors, neutrophil activation, and platelet activation have also been demonstrated in preeclampsia and are consistent with endothelial dysfunction.24 Inflammatory cytokines are known to be potent activators of the vascular endothelium and have been proposed as mediators of endothelial dysfunction during preeclampsia.25 Both tumor necrosis factor α (TNFα) and interleukin 1 β (IL-1β), interleukin-10 (IL-10) induce functional alterations in endothelial cells.26 Although the association of these inflammatory cytokines with the development of pre-eclampsia (PE) is generally assumed, the actual mechanism, and modes of dysregulation are still in strong debate. In two authoritative journal, the authors described a dysregulation of cytokine expression occurs in the pre-eclamptic placenta, with overexpression of IL-10 mRNA in placenta tissues and elevated plasma level (Am J Obstet Gynecol 1999;181:915-20; Obstet Gynecol 2002;100:327-31).27,28 In contrast, another influential journal describes deficiency in plasma production of IL-10 and decreasing plasma level of IL-10 (J Immunology, 1999, 163: 3491-5)29. Authors also measured the IL-10 released by in vitro culture of CTB from PE patients. The results also shows significantly alternation in IL-10 release by in vitro culture of PE CTB (Cytokine 23 2003;23:119-25)30.

We believed that studying the CTB itself is not enough to explain the pathogenesis of preeclampsia. CTB itself, and also the implantation environment are also expressed IL-10 and other inflammatory cytokines. We suggest assess the in situ specimen including placenta tissues and placental bed biopsies may include both the influence of CTB and its implantation environment. Besides, if IL-10 does play a role in the pathogenesis of preeclampsia, altering the expression IL-10 level may restore the PE phenotype to normal behavior. This is our purpose of observation in the following study.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia

Exclusion Criteria:

* no

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnacnt women
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-01; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Pan-Chyr, Study Chair — National Taiwan University Hospital Research Ethics Committee
Locations (1):
- Shih Jin-Chung, Taipei, Taiwan